CLINICAL TRIAL: NCT03072589
Title: A Phase 1 Open Label Study to Evaluate Adenosine 2A Receptor Agonist (Regadenoson) in Patients Undergoing Lung Transplantation
Brief Title: Study to Evaluate Adenosine 2A Receptor Agonist (Regadenoson) in Patients Undergoing Lung Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christine Lau, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Christine Lau, MD, Surgeon-in-Chief, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UVA-LAU-01; 1R01HL128492-01A1 (NIH)
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lung Transplant

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regadenoson infusion (Experimental): Dose escalation of Regadenoson infusion
  Interventions: Drug: Regadenoson infusion

INTERVENTIONS:
Drug: Regadenoson infusion — Dose escalation of Regadenoson when given as an infusion

SUMMARY:
This study will evaluate the maximum safe dose and duration of regadenoson (Lexiscan) that can be given to people who are having a lung transplant. Regadenoson will be given as a continuous IV infusion. All participants in the study will receive a regadenoson infusion beginning in the operating room during the lung transplant procedure. Participants will be assigned a certain dose of regadenoson to be given over a 12 or 24 hour period.

DETAILED DESCRIPTION:
Lung transplantation currently is one way to treat a variety of serious diseases and conditions such as emphysema, pulmonary fibrosis, and cystic fibrosis. Ischemia Reperfusion Injury (IRI) is a known problem that can happen during the first few days after a lung transplant. IRI can cause swelling of the lungs and low levels of oxygen. The most serious type of IRI can cause the transplanted lung to not work properly, it can even cause death. While new treatments and practices have been put into place to lower the chances of IRI, it is still a difficult problem to overcome after a lung transplant.

Medicines called Adenosine 2A receptors (A2AR) have been studied in animals with IRI for many years. Some of these studies suggest that with the use of A2AR medicines, the chance of IRI may be lowered or prevented. Regadenoson is an A2AR drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing a bilateral lung transplantation for end-stage lung disease and thus meet all criteria to be listed
* Male or female subject, 18 -75 years of age
* Subjects must sign a study specific informed consent prior to study entry
* Subjects must meet all of the following laboratory values:

  1. hemoglobin ≥ 6 g/dL,
  2. platelets > 75,000/mcL,
  3. aspartate aminotransferase (AST/SGOT)/ alanine aminotransferase (ALT /SGPT) < 2.5 X institutional upper limit of normal,
  4. serum creatinine < 1.5 mg/dL,
  5. INR < 1.5, PTT < 40 seconds

Exclusion Criteria:

* Subject requires preoperative extracorporeal membrane oxygenation (ECMO)
* Subject has second degree (Mobitz type I or II) or third-degree AV block or sinus node dysfunction
* Subject has history of a bleeding diathesis
* Subject has a history of clinically overt stroke within the past 3 years
* Subject has a history of severe hypertension not adequately controlled with anti-hypertensive medications (Systolic blood pressure ≥ 200 mmHg and/or Diastolic blood pressure ≥ 110 mmHg)
* Subjects who are receiving chronic anti-coagulation or anti-platelet therapy that would preclude surgery (prophylactic aspirin is acceptable)
* Subjects with a history of metastatic cancer
* Subjects with a history of seizure disorder
* Subjects who are receiving or have received within 30 days any other investigational agents
* Subjects who have received theophylline or aminophylline within 12 hours of study dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient tolerability of assigned dose and duration | Day 7
  Absence of a dose-limiting toxicity

SECONDARY OUTCOMES:
Activation of iNKT cells | 24 hours
  Activation of iNKT cells
Clinical Pulmonary Graft Dysfunction (PGD) score | 72 hours
  Evaluate for ischemia reperfusion injury
Inflammatory Cytokines in blood and bronchioalveolar lavage | 24 hours
  Inflammatory Cytokines in blood and bronchioalveolar lavage

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lau, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau CL, Beller JP, Boys JA, Zhao Y, Phillips J, Cosner M, Conaway MR, Petroni G, Charles EJ, Mehaffey JH, Mannem HC, Kron IL, Krupnick AS, Linden J. Adenosine A2A receptor agonist (regadenoson) in human lung transplantation. J Heart Lung Transplant. 2020 Jun;39(6):563-570. doi: 10.1016/j.healun.2020.02.003. Epub 2020 Feb 13. PMID 32503727